CLINICAL TRIAL: NCT00526175
Title: LAL-BR/2001: Study Treatment to Low Risk ALL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAL-BR/2001
Record Dates: First submitted 2007-09-06; First posted 2007-09-10 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Acute Lymphoblastic Leukemia; Minimal Residual Disease
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — Prednisone; Vincristine; Daunorubicin; Asparaginase; Cyclophosphamide; Methotrexate; Cytarabine; Mercaptopurine; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Prednisone — 60 mg/m2 day, i.v. or oral, dyas 1 to 27 30 mg/m2 day, i.v. or oral, days 28 to 35
Drug: Vincristine — 1,5 mg/m2 i.v., days 8, 15, 22 and 28
Drug: Daunorubicin — 30 mg/m2, i.v., days 8 and 15
Drug: L-Asparaginase — 10.000 UI/m2, i.m. or i.v., days 9 to 11, 16 to 18 and 23 to 25. Total: 9 doses.
Drug: Cyclophosphamide — 1000 mg/m2, i.v., day 22.
Drug: Methotrexate — Age <1 year 1-2 years 2-3 years > 3 years MTX 5 mg 8 mg 10 mg 12 mg
Drug: Cytosine Arabinoside — Edad <1 year 1-2 years 2-3 years > 3 years ARA-C 16 mg 16 mg 20 mg 30 mg
Drug: Mercaptopurine — 50 mg/m2,oral, days 1 to 7, 28-35 and 56-63
Drug: VP-16 — 150 mg/m2 i.v., days 14-15 and 42-43

SUMMARY:
The purpose of this study is increase the efficacy of consolidation (C1) after an intensification phase with high dose of methotrexate, applying analysis of minimal residual disease

DETAILED DESCRIPTION:
REMISION INDUCTION

Systemic chemotherapy:

Prednisolone (PDN):

* 60 mg/m2 day, i.v. or p.o., days 1 to 27
* 30 mg/m2 day, i.v. or p.o., days 28 to 35

Vincristine (VCR): 1,5 mg/m2 i.v., days 8, 15, 22 and 28. Daunorubicin (DNR): 30 mg/m2, i.v., days 8 and 15. L-asparaginase (L-ASA): 10.000 UI/m2, i.m. or i.v., days 9 to 11, 16 to 18 and 23 to 25.

Cyclophosphamide (CFM): 1000 mg/m2, i.v., day 22.

Intracranial chemotherapy

Methotrexate (MTX), cytosine (ARA-C) and hydrocortisone, days 1 and 22

CONSOLIDATION TREATMENT (WEEKS 6 TO 14)with INTENSIFICACIÓN (C-1)

* Mercaptopurine (MP) 50 mg/m2, p.o., days 1-7, 28-35 and 56-63
* MTX: 3g/m2, i.v., in 24 hours, days 1, 28 and 56.
* VP-16: 150 mg/m2 i.v., days 14-15 and 42-43
* ARA-C: 1000 mg/m2 i.v., in 3 hours, days 14-15 and 42-43
* Intrathecal treatment, days 1, 28 and 56.

REINDUCTION-CONSOLIDATION TREATMENT (R-C) (WEEKS 15 TO 23)

Dexamethasone (DXM):

* 6 mg/m2 day, p.o., days 1-21
* 3 mg/m2 day, p.o. or i.v., days 22-28 VCR: 1,5 mg/m2, i.v., days 1, 8 and 15 DNR: 30 mg/m2, i.v., days 1 and 8 L-ASA: 10.000 UI/m2 i.m. or i.v., days 8 and 9, 15 and 16, 22 and 23. CFM 1000 mg/m2 day, i.v., day 22 Mercaptopurine (MP) 50 mg/m2, p.o., days 35-42 MTX: 3g/m2, i.v., in 24 hours, day 35. VP-16: 150 mg/m2 i.v., days 49-50 ARA-C: 1.000 mg/m2 i.v., in 3 hours, days 49-50 Intrathecal treatment days 1 and 35.

MAINTENANCE TREATMENT (M-1)

Continuous treatment

* MP 50 mg/m2/day, p.o.
* MTX 20 mg/m2/week, i.m.

Reinductions

* VCR: 1,5 mg/m2 i.v., day 1.
* PDN: 30 mg/m2/day, i.v. or p.o., days 1 to 7
* L-ASA: 20.000 UI/m2, i.m. or i.v., day 1.
* Intrathecal treatment day 1 Five cycles, weeks 24, 30, 36, 42 and 48. During the week of administration cycle, continuous chemotherapy should be suspended.

Intrathecal treatment: At the start of any reinduction cycle

MAINTENANCE TREATMENT (M-2) (WEEKS 55-108)

* MP 50 mg/m2/day, p.o.
* MTX 20 mg/m2/week, i.m.
* Intrathecal treatment, weeks 54 and 108

At the end of treatment should be done the study of MRD (flux cytometry)

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of low risk acute lymphoblastic leukemia in children no treated previously

Exclusion Criteria:

* Mature B-ALL (FABL3) or with cytogenetic ALL "Burkitt-like" alterations (t[8;14], t[2;8], t[8;22])
* Mixed forms of ALL
* Acute Leukemia no differentiate
* Patients with coronary disorders, valvular or hypertensive cardiopathy
* Patients with chronic liver disorders
* Chronic pulmonary disorders
* Renal insufficiency
* Neurologic disfunctions
* ECOG 3 and 4
* No signed consent form

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2001-06; Primary Completion 2015-05 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of treatment in order to response rate, relapse free survival and global survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ribera Josep Mª, Dr, Study Chair — Germans Trias i Pujol Hospital; Bastida Pilar, Dr, Study Chair — Hospital Materno-Infantil Vall d'Hebron
Locations (25):
- Spain (25):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Valle Hebrón-Materno Infantil, Barcelona, Barcelona
  - Complejo Hospitalario Reina Sofía, Córdoba, Córdoba
  - Hospital Clínico San Carlos de Madrid, Madrid, Madrid
  - . Hospital Clínico Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Joan XXIII, Tarragona, Tarragona
  - Hospital Clínic, Valencia, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia, Valencia
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital de Badalona Germans Trias i Pujol, Badalona
  - Hospital de Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Basurtuko Ospitalea, Basurto
  - Hospital General de Guadalajara, Guadalajara
  - Complejo Hospitalario León, León
  - Complejo Asistencial Son Dureta, Palma de Mallorca
  - Hospital Clinico Universitario, Salamanca
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - H.U. Virgen del Rocio, Seville
  - Hospital Arnau de Vilanova, Valencia
  - Hospital Clínico de Valladolid, Valladolid

REFERENCES:
- See also: Spanish association of Haematology — http://www.aehh.org